CLINICAL TRIAL: NCT03135561
Title: A Pedometer-based Walking Intervention With and Without Email Counselling in General Practice: a Pilot Randomised Controlled Trial
Brief Title: A Pedometer-based Intervention With and Without Email Counselling in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Tomáš Větrovský, PhD Student, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pedometer-plus-email
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Physical Activity; Primary Care; General Practice
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pedometer-plus-email (Experimental)
  Interventions: Behavioral: pedometer-plus-email
- pedometer-only (Active Comparator)
  Interventions: Behavioral: pedometer-only

INTERVENTIONS:
Behavioral: pedometer-plus-email — After randomisation, participants will receive a pedometer and will be instructed to wear the pedometer daily for the next four months, check the step count every evening and gradually increase their daily number of steps to at least 10,000. They will also be required to upload data to a website at least once a week. During the intervention period, patients will receive 8 counselling emails based on behavioural techniques.
  Arms: pedometer-plus-email
Behavioral: pedometer-only — After randomisation, participants will receive a pedometer and will be instructed to wear the pedometer daily for the next four months, check the step count every evening and gradually increase their daily number of steps to at least 10,000. They will also be required to upload data to a website at least once a week. There will be no further interaction during the intervention period unless they fail to upload data, in which case they will be offered technical support.
  Arms: pedometer-only

SUMMARY:
A two-arm parallel randomised controlled trial comparing pedometer-based intervention with and without email counselling in a primary care setting. Physically inactive patients from four general practices will be randomised to the pedometer-plus-email group or to the pedometer-alone group. All patients will be instructed to gradually increase the daily number of steps to at least 10,000. Patients in the pedometer-plus-email group will receive 8 counselling emails based on behavioural techniques. The primary outcome will be change in average daily steps measured during 7-day period at baseline and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* physically inactive, i.e. takes less than 8,000 steps per day at baseline
* registered at the participating general practice,
* over 18 years of age,
* regular email user, and willing to use email for the purpose of the study,
* has a home computer with access to the Internet.

Exclusion Criteria:

* medical or psychiatric condition which the general practitioner considers as inappropriate for participating in the intervention (e.g., terminal illness, psychotic illness, chronic disorders or diseases that seriously influence the ability to be physically active, dementia or significant cognitive impairment, unable to move about independently),
* medical, personal of family condition which the general practitioner considers temporarily affects mean daily step count at baseline (e.g., acute illness, holiday or business trip),
* pregnant woman,
* currently engaging in regular sports or exercise (at least twice a week),
* failure to upload pedometer data to a website at baseline assessment,
* failure to give informed consent with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
average daily step count | 12 weeks
  change in average daily steps measured during 7-day period at baseline and at 12 weeks

SECONDARY OUTCOMES:
body weight | 12 weeks
  measured to the nearest kg
systolic blood pressure | 12 weeks
  measured to the nearest mmHg
diastolic blood pressure | 12 weeks
  measured to the nearest mmHg
waist circumference | 12 weeks
  recorded with a measurement tape to the nearest cm
hip circumference | 12 weeks
  recorded with a measurement tape to the nearest cm

OTHER OUTCOMES:
health-related quality of life | 12 weeks
  assessed with the 36-Item Short Form Health Survey (SF-36)
anxiety | 12 weeks
  assessed with the anxiety subscale of the Hospital Anxiety and Depression Scale
depression | 12 weeks
  assessed with the depression subscale of the Hospital Anxiety and Depression Scale
self-efficacy | 12 weeks
  assessed with the Czech version of the General Self-Efficacy scale

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Vetrovsky, MD, Principal Investigator — Charles University, Czech Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vetrovsky T, Cupka J, Dudek M, Kuthanova B, Vetrovska K, Capek V, Bunc V. A pedometer-based walking intervention with and without email counseling in general practice: a pilot randomized controlled trial. BMC Public Health. 2018 May 16;18(1):635. doi: 10.1186/s12889-018-5520-8. PMID 29769107